CLINICAL TRIAL: NCT04925622
Title: Complex Eye Movements in Parkinson's Disease and Related Movement Disorders
Status: Completed | Type: Observational
Sponsor: Saccadous, Inc. (Other)
Collaborators: Dignity Health (Other); Barrow Neurological Institute (Other)
Responsible Party: Sponsor
Other Study IDs: SACCADOUSPDPH1
Record Dates: First submitted 2021-06-01; First posted 2021-06-14 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2022-05

CONDITIONS: Parkinson Disease; Parkinson's Disease and Parkinsonism; Progressive Supranuclear Palsy; Corticobasal Degeneration; Parkinsonian Disorders; Essential Tremor; Vascular Parkinsonism; Multiple System Atrophy, Parkinson Variant; Parkinsonian Syndrome; Huntington Disease
Keywords: Eye Movement; Neurological Diagnosis; Saccades; Microsaccades
MeSH Terms: conditions — Parkinson Disease; Parkinsonian Disorders; Supranuclear Palsy, Progressive; Corticobasal Degeneration; Essential Tremor; Multiple System Atrophy; Huntington Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (3):
- Control: No symptoms of neurological condition
  Interventions: Diagnostic Test: Complex eye movement exam
- Parkinson's disease: Parkinson's disease diagnosis
  Interventions: Diagnostic Test: Complex eye movement exam
- Non-PD Movement disorder: Non-PD with other movement disorder such as progressive supranuclear palsy, multiple system atrophy, essential tremor, corticobasal degeneration, vascular Parkinsonism, or Parkinsonian syndromes
  Interventions: Diagnostic Test: Complex eye movement exam

INTERVENTIONS:
Diagnostic Test: Complex eye movement exam — Subjects will undergo a complex eye exam which will capture fixation, optokinetic nystagmus, guided saccades, microsaccades, smooth pursuit, and pupillometry.
  Eye tracking equipment will be set and calibrated to the participant who will then perform the full 10 minute testing protocol with instructions from the investigator. After this, they will take a five minute break. The oculomotor testing protocol will be repeated twice.

SUMMARY:
Diagnosing Parkinson's disease (PD) depends on the clinical history of the patient and the patient's response to specific treatments such as levodopa. Unfortunately, a definitive diagnosis of PD is still limited to post-mortem evaluation of brain tissues. Furthermore, diagnosis of idiopathic PD is even more challenging because symptoms of PD overlap with symptoms of other conditions such as essential tremor (ET) or Parkinsonian syndromes (PSs) such as progressive supranuclear palsy (PSP), multiple system atrophy (MSA), corticobasal degeneration (CBD), or vascular Parkinsonism (VaP). Based on the principle that PD and PSs affect brain areas involved in eye movement control, this trial will utilize a platform that records complex eye movements and use a proprietary algorithm to characterize PSs. Preliminary data demonstrate that by monitoring oculomotor alterations, the process can assign PD-specific oculomotor patterns, which have the potential to serve as a diagnostic tool for PD.

This study will evaluate capabilities of the process and its ability to differentiate PD from other PSs with statistical significance. The specific aims of this proposal are: To optimize the detection and analysis algorithms, and then to evaluate the process against neurological diagnoses of PD patients in a clinical study.

DETAILED DESCRIPTION:
In the Phase I, complex eye movements, including Fixation, Optokinetic Nystagmus (OKN), Guided Saccades, Microsaccades, Smooth Pursuit, and Pupillometry will be measured in 90 subjects (30 PD, 30 non-PD with other movement disorders (PSP, ET, CBD, etc.), and 30 normal defined as not having any symptoms of any neurological condition.) The patients will be classified according to clinical evaluations and clinical follow ups performed by Dr. Holly Shill, Director of the Lonnie and Muhammad Ali Parkinson Center at the Barrow Neurological Institute (Phoenix, AZ). A 3-way analysis will be performed to troubleshoot and optimize the detection and classification algorithms. At this stage, these results will only be used for the evaluation of the diagnostic capability of the tool and not to treat or diagnose the patient. The product is portable with the potential to be an accurate tool to diagnose PD. This tool will provide substantial support to neurologists by validating or complementing the clinical tests currently used to diagnose PD. Successful diagnosis of PD can open new avenues for diagnosing other neurological conditions.

ELIGIBILITY:
Inclusion Criteria:

* Patients assigned to PD or non-PD group based on medical records
* Control participants will be without previous diagnosis of a movement disorder
* Experimental groups and normal controls matched by age and gender

Exclusion Criteria:

* Severe drug/alcohol use
* Severe medical problems (e.g. terminal cancer)
* Macular degeneration
* Inability to consent
* Patients at 4 or more on the Hoehn-Yahr scale
* Inability to complete experimental protocol

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Both male and females eligible; control group will be age and gender matched
Study Population: Community Sample
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2021-01-04 (Actual); Primary Completion 2022-04-15 (Actual); Study Completion 2022-04-15 (Actual)

PRIMARY OUTCOMES:
Percent of patients accurately diagnosed with SaccadeDX | One test (approx. 1 hour)
  The primary outcome measure will be accurate diagnosis in over 75% of patients; accuracy will be determined with statistical significance.
  Each eye movement test will produce a unique signature. Using a historical database and machine learning, the SaccadeDX algorithm will match the signature to a specific patient group (PD, non-PD movement disorder, control) resulting in a "SaccadeDX diagnosis". Once the patients are fully enrolled, the SaccadeDX diagnosis will be compared to the diagnosis previously made by the sub-investigator. Accurate diagnosis will be defined as a SaccadeDX diagnosis that matches the initial diagnosis provided by the sub-investigator.

CONTACTS AND LOCATIONS:
Overall Officials: Hector Rieiro, PhD, Principal Investigator — Saccadous Chief Technology Officer
Locations (1):
- Dignity Health / St. Joseph's Hospital and Medical Center, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No
Proprietary and competitive data